CLINICAL TRIAL: NCT01074827
Title: Strength Training or Treadmill Walking? A Randomized Control Study on the Effect on Gait in Multiple Sclerosis
Brief Title: Improving Gait in Multiple Sclerosis (MS) - Strength Training or Treadmill Walking?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Helse Midt-Norge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/225
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Walking ability; Strength; Balance; Treadmill walking
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treadmill group (Experimental): Specific gait training on treadmill
  Interventions: Other: Strength training and treadmill training
- Strength training group (Experimental): Eight weeks of intensive strength training
  Interventions: Other: Strength training and treadmill training

INTERVENTIONS:
Other: Strength training and treadmill training — Eight weeks of intensive strength training or treadmill training

SUMMARY:
The objective of this study is to evaluate the effect of strength training for the lower extremities and treadmill training on walking ability in persons with Multiple Sclerosis. The study is a randomized control trial with two groups and the intervention is 8 weeks of intensive strength training or treadmill walking. Primary outcome measure is walking ability, secondary outcome measures are balance, work economy and strength.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Multiple Sclerosis,classified as relapsing remitting,or primary/secondary progressive
* Expanded Disability Status Scale (EDSS)score of ≤ 6
* Reduced walking ability (subjectively experienced)

Exclusion Criteria:

* persons with a level of ataxia, clinically assessed, that would affect their ability to perform the training.
* spasticity requiring stretching og treatment with baclofen.
* Other, not MS-related, conditions affecting walking ability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Walking ability | 8 weeks

SECONDARY OUTCOMES:
Strength | 8 weeks
Work economy O2 | 8 weeks
Balance | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Siri M, Brændvik, Study Chair — St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Braendvik SM, Koret T, Helbostad JL, Loras H, Brathen G, Hovdal HO, Aamot IL. Treadmill Training or Progressive Strength Training to Improve Walking in People with Multiple Sclerosis? A Randomized Parallel Group Trial. Physiother Res Int. 2016 Dec;21(4):228-236. doi: 10.1002/pri.1636. Epub 2015 Jun 25. PMID 26110230